CLINICAL TRIAL: NCT05938036
Title: PUERTA: A P2A Multi-center, Randomized, Double-blind, Placebo-controlled Study Assessing Safety and Efficacy of the eNAMPT Targeting mAb ALT-100 in Moderate/Severe ARDS/VILI Patients
Brief Title: Study of Safety and Efficacy of ALT-100mAb in Participants With Moderate/Severe ARDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aqualung Therapeutics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-100-002
Record Dates: First submitted 2023-05-17; First posted 2023-07-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A : ALT-100 mAB (Dose Escalation) (Experimental): 90 eligible participants will be randomized at a 2:1 ratio to receive a single dose of ALT-100 mAb.
  Part A will assess 2 doses of ALT-100 mAb in sequentially enrolled cohorts of up to 9 participants in each cohort. (Randomised, Double-blind) Drug: ALT-100 mAb Dosage Form: Sterile liquid, pH 5.5, Dosage: 0.4 mg/kg (Cohort 1a) and 1.0 mg/kg (Cohort 2a) Dosage Form & Route of Admin: Solution for IV Infusion
  Interventions: Drug: ALT-100 mAb
- Part A Placebo (Placebo Comparator): Part A participants with acute respiratory distress syndrome (ARDS) (Randomised, Double-blind) Dosage Form & Route of Admin: Normal Saline Solution for IV Infusion
  Interventions: Drug: ALT-100 (Placebo)
- Part B (Dose Expansion) ALT-100 mAb (Experimental): Approximately 9 participants in each cohort in Part A, additional participants (up to 36 per dose cohort) may be enrolled into 2 dose expansion cohorts, the dose of which will be determined by the SRC. Drug: AT-02 Dosage: Will be decided by the SCR Route of Admin: Solution for IV Infusion
  Interventions: Drug: ALT-100 mAb

INTERVENTIONS:
Drug: ALT-100 mAb — Experimental: Part A : ALT-100 mAB (Dose Escalation) 90 eligible participants will be randomized at a 2:1 ratio to receive a single dose of ALT-100 mAb.
  Arms: Part A : ALT-100 mAB (Dose Escalation); Part B (Dose Expansion) ALT-100 mAb
Drug: ALT-100 (Placebo) — Normal saline solution via IV solution
  Arms: Part A Placebo

SUMMARY:
A Phase 2a, multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of ALT-100mAb in patients with moderate to severe ARDS.

DETAILED DESCRIPTION:
PUERTA is a Phase 2a, randomized, double-blind, placebo-controlled study in adults with moderate to severe ARDS consequent to sepsis, septic shock, trauma, and/or bacterial or viral pneumonia who have been hospitalized. The safety and tolerability, PK, preliminary efficacy, and PD of a single infusion of ALT-100 mAb will be assessed. All participants will receive study drug within 12 hours of their ARDS diagnosis and within 4 hours of initiation of MV (mechanical ventilation).

It is planned that 90 eligible participants will be randomized at a 2:1 ratio to receive a single dose of either ALT-100 mAb or placebo via IV infusion at the time the diagnosis of moderate to severe ARDS is confirmed. An additional 9 participants may be randomized if an optional cohort of low or intermediate ALT-100 mAb dose is enrolled.

The study will be conducted in 2 parts:

* Part A: a dose escalation phase followed by
* Part B: dose expansion phase

Dose Escalation (Part A) Part A will assess 2 doses of ALT-100 mAb in sequentially enrolled cohorts of up to 9 participants in each cohort. The planned doses of ALT-100 mAb are 0.4 mg/kg (Cohort 1a) and 1.0 mg/kg (Cohort 2a).

Dose Expansion (Part B) Following SRC review of all data up to Day 29 from the 9 participants in each cohort in Part A, additional participants (up to 36 per dose cohort) may be enrolled into 2 dose expansion cohorts, the dose of which will be determined by the SRC. Part B will further explore the safety, preliminary efficacy, PK, and systemic biomarker profile of ALT-100 mAb.

Participants enrolled in Part A may not be re-enrolled in Part B.

The screening, Treatment, and Safety Follow-up schedules are the same for Part A (dose escalation) and Part B (dose expansion) cohorts.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a participant must meet all of the following criteria:

1. Hospitalized (or documentation of a plan to admit to the hospital if the patient is in an emergency department) male or non-pregnant female 18 years and above of age at time of enrollment.
2. Participant (or LAR) is able and willing to provide written informed consent, which includes compliance with study requirements and restrictions listed in the consent form.
3. Participant has a diagnosis of moderate or severe ARDS:

   A participant with a diagnosis of moderate or severe ARDS according to the Berlin definition of ARDS:
   1. Acute onset of respiratory failure within 1 week of a known clinical insult or new or worsening respiratory symptoms.
   2. Respiratory failure associated with known ARDS risk factors and not fully explained by either cardiac failure or fluid overload (an objective assessment of cardiac failure or fluid overload is needed if no risk factors for ARDS are present).
   3. Radiological abnormalities on chest x-ray or computed tomography (CT) scan, ie, bilateral opacities that are not fully explained by effusions, nodules, masses, or lobar/lung collapse.
   4. Hypoxemia:

   i. Moderate ARDS: PaO2/FiO2 more than 100 mmHg (more than 13.3 kPa) to 200 mmHg and below (26.6 kPa and below) with PEEP 5 cmH2O and above, or imputed SpO2/FiO2 equivalent.

   ii. Severe ARDS: PaO2/FiO2 100 mmHg and below (13.3 kPa and below) with PEEP 5 cmH2O and above.

   OR Participant presents with acute respiratory failure phenotypically similar to ARDS in a setting demonstrating clinical risk for ARDS, whether or not they meet the Berlin criteria, and requiring heated and humidified HFNC 30 L/min and above and 100 percent FiO2, or NIPPV (ie, BiPAP/CPAP) for hypoxemia.

   OR Participant presents with acute respiratory failure phenotypically similar to ARDS in a setting demonstrating clinical risk for ARDS, do not meet the Berlin criteria, and initially treated with 12 continuous hours and above with HFNO using gas flow of 40 L/min and above or treated with non-invasive ventilation (NIV), and has a PEEP of 5 cm and above H2O and PaO2/FIO2 below 300 mm Hg.
4. Administration of study treatment must be planned to occur within 12 hours of the participant's moderate or severe ARDS diagnosis and within 4 hours of initiation of MV (in the case of individuals requiring immediate MV).
5. Females must be non-pregnant and non-lactating, and either surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use highly effective contraceptive method (oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones, a vaginal ring or an intrauterine device [IUD]) from screening until study completion or be post-menopausal for 12 months and above. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels at screening for amenorrheic female participants, but the result is not required prior to enrollment. Female participants whose only partner has had a vasectomy, and female participants who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible for participation.
6. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and admission and be willing to have additional pregnancy tests as required throughout the study.
7. Males must be surgically sterile (more than 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP his partner must be surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from screening until study completion, including the Follow-up Period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner (WOCBP) that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Male participants whose female partner is post-menopausal, and participants who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible.
8. Male participants must agree to refrain from donating sperm from screening until study completion, including the Follow-up Period, for at least 60 days after the last dose of study treatment.
9. Participant is willing and able to undergo all study procedures and attend the scheduled follow-up visit/s per protocol.

Exclusion Criteria:

A participant who meets any of the following criteria must be excluded from the study:

1. Participants with ARDS consequent to COVID-19 infection.
2. Participants requiring immediate MV who have been intubated and on MV for more than 4 hours prior to the planned administration of study treatment on Day 1
3. Moribund participant not expected to survive more 24 hours, in the opinion of the Investigator.
4. Use of extracorporeal life support (eg, ECMO) or, in the opinion of the Investigator, there is a high likelihood that extracorporeal life support will be initiated within 48 hours after randomization.
5. Participant has an underlying clinical condition where, in the opinion of the Investigator, it would be unlikely that the participant would be able to come off ventilation, eg, chronic progressive neuromuscular or respiratory disease.
6. Severe chronic respiratory disease (eg, known chronic obstructive pulmonary disease [COPD], pulmonary arterial hypertension [PAH], idiopathic pulmonary fibrosis [IPF], interstitial lung disease [ILD]) requiring supplemental oxygen therapy or MV pre-hospitalization (eg, prior to ARDS diagnosis).
7. Evidence of life-threatening dysrhythmia (eg, ventricular tachycardia, ventricular fibrillation) or cardiac arrest on presentation.
8. Evidence of new or preexisting decompensated heart failure.
9. Absolute neutrophil count lesser than1000 per mm3.
10. Platelet count less than 50000 per mm3.
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 5 × ULN.
12. Estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73m2 (based on MDRD equation) or requiring hemofiltration or dialysis.
13. Known or suspected active and untreated tuberculosis (TB), HIV, hepatitis B or C infection.

    Note: Results of TB, hepatitis B and C, and HIV tests are not required prior to enrollment if there is no suspicion of active infection.
14. Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies, fusion proteins, ALT-100 excipients, or a history of drug or other allergy including severe allergic reaction that in the opinion of the Investigator or MM, contraindicates participant participation.
15. Use of any immunomodulatory biologic (eg, anti-IL-1, anti-IL-6R, anti-TNF, inhibitors of complement signaling), cell therapies (eg, mesenchymal stem cells), or small molecule Janus kinase (JAK) inhibitors within the past 7 days or within 5 half-lives (whichever is longer), or planned use of any of these agents from screening until Day 60 of the study, unless approved by the MM. The following will be allowed/ disallowed as indicated:

    1. Immunomodulatory biologics for treatment of COVID-19 are excluded and should not be used until Day 60 unless discussed with the MM. Other non-biologic immunomodulators (non-JAK inhibitors), eg, medicines for previous transplantation, or DMARDS, if on a stable dose for 8 weeks and above are permitted.
    2. Ongoing chronic (4 weeks and above) use of corticosteroids more than 10 mg/day of prednisone or equivalent at the time of randomization is prohibited. A corticosteroid dose that has been tapered to 10 mg or less within 14 days of randomization is also prohibited.
16. Participants who have circulatory shock requiring vasopressors at randomization or within 24 hours prior to randomization will be excluded from study participation.

    Participants who present at screening with ARDS and septic shock may be enrolled if the participant is on one vasopressor or, if on 2 vasopressors, if the Levofed (norepinephrine) dose is 1 microgram/kg/min and lesser.

    Participants with ARDS and septic shock who are on 3 and above vasopressors ie, Vasopressin, Levofed (norepinephrine), Neosynephrine (phenelephreine), at screening are excluded from study participation.

    Participants with ARDS and septic shock who are on 2 vasopressors where the Levofed dose is more than 1 micro gram/kg/min are excluded from study participation.
17. Participation in a clinical research study evaluating another IP or therapy within 3 months and less than 5 half-lives of the IP prior to the Screening Visit.
18. Any physical examination findings, and/or history of any other illness, concomitant medications, or recent live vaccines that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
19. Administered a live vaccine within 14 days prior to IP administration and throughout the duration of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Safety and tolerability of a single intravenously (IV) infused dose of ALT-100 in participants with moderate to severe ARDS: Incidence and severity of treatment-emergent adverse events (TEAEs) from Day 1 to end of study (EOS). | Up to 60 days
  Assessment will be done by measuring the following parameter:
  • Incidence and severity of treatment-emergent adverse events (TEAEs) from Day 1 to end of study (EOS).

SECONDARY OUTCOMES:
To evaluate the impact of a single IV infusion of ALT-100 on respiratory support. | Up to 29 Days
  Assessment will be done by measuring Number of Mechanical Ventilation-free days (MVFD) over 28 days following study treatment (ie, MVFDs by Day 29).
To assess the effect of ALT-100 on duration of hospitalization: Time to hospital discharge based on days since admission to discharge. | Up to 29 Days
  Assessments will be done by:
  - Time to hospital discharge based on days since admission to discharge.
To assess the effect of ALT-100 on duration of hospitalization: Hospital Free Days (HFD) to Day 29. | Up to 29 Days
  Assessments will be done by:
  - Hospital Free Days (HFD) to Day 29.
To assess the effect of ALT-100mAb as measured by the Sequential Organ Failure Assessment (SOFA) score. | Up to 29 Days
  Assessments will be done by:
  - Total and component Sequential Organ Failure Assessment (SOFA) score assessed daily while in the intensive care unit (ICU).
  The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Score ranges from 0 (best) to 24 (worst) points
To assess the effect of ALT-100 mAb on oxygen-related parameters :Changes as measured by change from baseline in plethysmographic pulse oximetry derived oxygen saturation / fraction of inspired oxygen and ROX Index | Up to 29 Days
  Assessments will be done by:
  • Changes as measured by change from baseline in plethysmographic pulse oximetry derived oxygen saturation / fraction of inspired oxygen (SpO2/FiO2) and ROX Index (SpO2/FiO2 divided by respiratory rate [RR]), assessed daily while hospitalized.
To assess the effect of ALT-100 mAb on oxygen-related parameters: If the participant is receiving MV, the P/F ratio will be used (ie, partial pressure of oxygen [PaO2]/FiO2). | Up to 29 Days
  Assessments will be done by:
  • If the participant is receiving MV, the P/F ratio will be used (ie, partial pressure of oxygen [PaO2]/FiO2).
To assess the effect of ALT-100 mAb on oxygenation requirements. | Up to 29 Days
  Assessments will be done by:
  - Incidence and duration of oxygen use (via conventional oxygen therapy, or non-invasive respiratory support positive pressure by face mask or HFNO) during the study.
To assess the effect of ALT-100 mAb on requirement for vasoactive support | Up to 29 Days
  Assessment will be done by:
  - Number of days of vasoactive agent usage Vasopressor free days
Pharmacodynamics : To investigate the effects of ALT-100 mAb on immune function biomarkers and cellular response. Changes from baseline in plasma levels of extracellular nicotinamide phosphoribosyl transferase and other biomarkers of interest. | Up to 29 Days
  To investigate the effects of ALT-100 mAb on immune function biomarkers and cellular response. Assessments will be done by:
  - Changes from baseline in plasma levels of extracellular nicotinamide phosphoribosyl transferase (eNAMPT) and other biomarkers of interest including but not limited to TNF-α, IL-1β, IL-1RA, IL-6, Angiopoietin-2.
Pharmacodynamics: To investigate the effects of ALT-100 mAb on immune function biomarkers and cellular response. Changes from baseline in cellular response with ALT-100 compared to placebo. | Up to 29 Days
  To investigate the effects of ALT-100 mAb on immune function biomarkers and cellular response. Assessments will be done by:
  - Changes from baseline in cellular response with ALT-100 compared to placebo, as assessed by: neutrophil, monocyte, and lymphocyte counts in whole blood.
Pharmacokinetics - To characterize the plasma PK profile of single IV infused doses of ALT-100 : Determination of plasma concentrations of ALT-100 mAb. | Up to 60 days
  To characterize the plasma PK profile of single IV infused doses of ALT-100. Assessment will be done to
  • Determination of plasma concentrations of ALT-100 mAb.
PK of single IV infused dose of ALT-100 | Up to 60 days
  Estimation of PK parameter
Number of participants with abnormal clinically significant clinical laboratory results | Up to 60 days
  Clinical laboratory tests include hematology, chemistry, coagulation and urinalysis.
Number of participants with abnormal clinical vital signs | Up to 60 days
  Vital signs include blood pressure, heart rate, respiration rate, body temperature
To further evaluate the safety and tolerability of a single intravenously(IV) infused dose of ALT-100 mAb through physical examination | Up to 60 days
  Secondary safety and tolerability outcomes while hospitalized or if discharged on Days 8, 15, 22, 29, and 60 will include:
  • Physical examination
Safety - To further evaluate the safety and tolerability of a single intravenously (IV) infused dose of ALT-100 mAb: Secondary safety and tolerability outcomes will include: Concomitant medication use | Up to 60 days
  Secondary safety and tolerability outcomes while hospitalized or if discharged on Days 8, 15, 22, 29, and 60 will include:
  • Concomitant medication use
Safety - To further evaluate the safety and tolerability of a single intravenously (IV) infused dose of ALT-100 mAb: Secondary safety and tolerability outcomes will include: Oxygenation (FiO2 and PaO2 or SpO2) | Up to 60 days
  Secondary safety and tolerability outcomes while hospitalized or if discharged on Days 8, 15, 22, 29, and 60 will include:
  • Oxygenation (FiO2 and PaO2 or SpO2)
Safety - To further evaluate the safety and tolerability of a single intravenously (IV) infused dose of ALT-100 mAb: Secondary safety and tolerability outcomes will include: Ventilation support. | Up to 60 days
  Secondary safety and tolerability outcomes while hospitalized or if discharged on Days 8, 15, 22, 29, and 60 will include:
  • Ventilation support: heated and humidified high flow nasal O2 [HFNO]
Safety - To investigate the presence of anti-ALT-100 mAb antibodies. | Up to 60 days
  To investigate the presence of anti-ALT-100 mAb antibodies.
  Assessment will be done by:
  Presence and characterization of ADA over the study period (baseline [Day 1 pre-dose], and post treatment on Days 8, 15, 29, and 60).

OTHER OUTCOMES:
Exploratory: detection of NAMPT genetic variants in blood: Determination of ARDS-associated NAMPT promoter SNP expression in baseline blood samples from all participants using a NAMPT genotyping platform. | Up to 60 days
  Exploratory detection of NAMPT genetic variants in blood
  Assessment will be done by:
  - Determination of ARDS-associated NAMPT promoter SNP expression in baseline blood samples from all participants using a NAMPT genotyping platform.
Exploratory: detection of NAMPT genetic variants in blood: Assessment of predictive capacity of NAMPT SNPs and plasma eNAMPT levels to identify participants who respond to single dose treatment with ALT-100 mAb. | Up to 60 days
  Exploratory detection of NAMPT genetic variants in blood
  Assessment will be done by:
  - Assessment of predictive capacity of NAMPT SNPs and plasma eNAMPT levels to identify participants who respond to single dose treatment with ALT-100 mAb.
Exploratory - To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care: Change from baseline in LIS (if performed) daily while hospitalized. | Up to 60 days
  To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care (eg, LIS, chest radiography, PaO2/FiO2, need for extracorporeal membrane oxygenation [ECMO])
  Assessments will be done by:
  - Change from baseline in LIS (if performed) daily while hospitalized.
Exploratory - To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care: Change from baseline in chest radiographic assessment (if performed). | Up to 60 days
  To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care (eg, LIS, chest radiography, PaO2/FiO2, need for extracorporeal membrane oxygenation [ECMO])
  Assessments will be done by:
  - Change from baseline in chest radiographic assessment (if performed).
Exploratory - To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care: Change from baseline in P/F ratio (if performed) daily while hospitalized. | Up to 60 days
  To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care (eg, LIS, chest radiography, PaO2/FiO2, need for extracorporeal membrane oxygenation [ECMO])
  Assessments will be done by:
  - Change from baseline in P/F ratio (if performed) daily while hospitalized.
Exploratory - To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care (eg, LIS, chest radiography, PaO2/FiO2, need for extracorporeal membrane oxygenation [ECMO]) Utilization of ECMO. | Up to 60 days
  To explore the effect of ALT-100 on other measurements of lung injury that may be performed during standard care (eg, LIS, chest radiography, PaO2/FiO2, need for extracorporeal membrane oxygenation [ECMO])
  Assessments will be done by:
  - Utilization of ECMO.
Exploratory - To assess the effect of ALT-100 on respiratory support requirements over time: MVFDs by Days 8, 15, 22, and 60. | Up to 60 days
  To assess the effect of ALT-100 on respiratory support requirements over time
  Assessment will be done by:
  - MVFDs by Days 8, 15, 22, and 60.
Exploratory - To assess the effect of ALT-100 on respiratory support requirements over time: Proportion of participants not on MV support on Days 8, 15, 22, 29, and 60. | Up to 60 days
  To assess the effect of ALT-100 on respiratory support requirements over time
  Assessment will be done by:
  - Proportion of participants not on MV support on Days 8, 15, 22, 29, and 60.
Exploratory - To assess the effect of ALT-100 on respiratory support requirements over time: Number of participants progressing from non-invasive to invasive MV by Days 8, 15, 22, 29, and 60. | Up to 60 days
  To assess the effect of ALT-100 on respiratory support requirements over time
  Assessment will be done by:
  - Number of participants progressing from non-invasive to invasive MV by Days 8, 15, 22, 29, and 60.
Exploratory - To assess the effect of ALT-100 on respiratory support requirements over time: Time of progression from non-invasive to invasive MV to Day 60. | Up to 60 days
  To assess the effect of ALT-100 on respiratory support requirements over time
  Assessment will be done by:
  - Time of progression from non-invasive to invasive MV to Day 60.
Exploratory - To assess the effect of ALT-100 on respiratory support requirements over time: Proportion of participants weaned from MV within 28-days from treatment (by Day 29). | Up to 60 days
  To assess the effect of ALT-100 on respiratory support requirements over time
  Assessment will be done by:
  - Proportion of participants weaned from MV within 28-days from treatment (by Day 29).
Exploratory - To explore the effect of ALT-100 mAb on mortality: Mortality in all participants by Days 8, 15, 22, 29, and 60. | Up to 60 days
  To explore the effect of ALT-100 mAb on mortality
  Mortality will be assessed by:
  - Mortality in all participants by Days 8, 15, 22, 29, and 60.
Exploratory - To explore the effect of ALT-100 mAb on mortality: Time to death by Day 60. | Up to 60 days
  To explore the effect of ALT-100 mAb on mortality
  Mortality will be assessed by:
  - Mortality in all participants by Days 8, 15, 22, 29, and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Stan Miele, Study Director — Aqualung Therapeutics Corp.
Locations (1):
- Banner University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not being shared with other researchers.